CLINICAL TRIAL: NCT04184791
Title: Computational Modeling of 60 Hz Subthalamic Nucleus Deep Brain Stimulation for Gait Disorder in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Ritesh Ramdhani, MD, Assistant Professor of Neurology, Northwell Health
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 19-0217; R21NS111301 (NIH)
Record Dates: First submitted 2019-11-22; First posted 2019-12-04 (Actual); Results first posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-02

CONDITIONS: Parkinson Disease
Keywords: Deep Brain Stimulation; Parkinson's Disease; Wearable Sensors
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Deep Brain Stimulation(DBS) OFF Medication (Experimental): Subthalamic-DBS in the Levodopa OFF state.
  Interventions: Device: Deep Brain Stimulation
- Deep Brain Stimulation(DBS) ON Medication (Experimental): Subthalamic-DBS in the Levodopa ON state.
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — Each DBS electrode contact will be reprogrammed in 60hz and High Frequency Stimulation (180hz) in the Levodopa ON (medicated) and OFF (unmedicated) conditions.

SUMMARY:
The objective of this study is to further the understanding and application of 60Hz subthalamic deep brain stimulation (STN-DBS) in Parkinson's patients with gait disorder. The investigators will achieve this through 2 study aims:

1. Determine the impact of 60Hz subthalamic deep brain stimulation on gait kinematics using wearable sensors
2. Develop machine learning models to predict optimal subthalamic deep brain stimulation frequency based on wearable sensors

DETAILED DESCRIPTION:
Gait disorder, which manifests as shuffling, reduction in speed, multistep turning, and/or freezing of gait (FOG), can arise later in the Parkinson's disease (PD) course and cause significant disability. Ultimately, patients are at risk for falls and can become socially isolated due to their mobility limitations. These symptoms tend not to respond to high frequency STN-DBS. However, lower frequency stimulation (60-80Hz) of the STN in treating gait disorder and/or freezing of gait has demonstrated benefit. This study potentially can expand knowledge of 60hz DBS while improving its utilization in combination with PD medications-enabling sustainable and possibly predictable therapeutic benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 21-80
2. Patients diagnosed with Parkinson's disease (PD)
3. PD subjects who have bilateral STN-DBS (greater than 3 months) or in the preoperative stage of being implanted with bilateral STN-DBS
4. Have underlying gait disorder
5. Currently treated with oral levodopa therapy
6. Willingness to comply with all study procedures

Exclusion Criteria:

1. Cognitive deficits based on historical record that limit participant compliance with study protocol
2. Vestibular disorder or musculoskeletal problems affecting gait or balance

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ritesh Ramdhani, MD, Principal Investigator — Northwell Health
Locations (1):
- Northwell Health, Great Neck, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All Subjects were recruited through the Movement Disorders Center at Northwell Health, NY.
Groups:
- Overall Study: 4 Phases: I - OFF DBS/OFF MED II- 180Hz DBS/ON MED III- 60Hz DBS/ON MED IV: OFF DBS/ON MED
Period: OFF Med/OFF DBS
Arm/Group | Overall Study
Started | 24
Completed | 22
Not Completed | 2
Period: 180Hz DBS ( OFF MED)
Arm/Group | Overall Study
Started | 24
Completed | 22
Not Completed | 2
Period: 180Hz (ON MED)
Arm/Group | Overall Study
Started | 24
Completed | 22
Not Completed | 2
Period: 60Hz DBS (OFF MED)
Arm/Group | Overall Study
Started | 24
Completed | 22
Not Completed | 2
Period: 60Hz (ON Med)
Arm/Group | Overall Study
Started | 24
Completed | 22
Not Completed | 2
Period: ON MED/OFF DBS
Arm/Group | Overall Study
Started | 24
Completed | 22
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Deep Brain Stimulation(DBS) OFF & ON Medication: Subthalamic-DBS in the Levodopa OFF and ON state.
  Deep Brain Stimulation: Each DBS electrode contact will be reprogrammed in 60hz and High Frequency Stimulation (180hz) in the OFF (unmedicated) and ON (medicated) conditions.
Arm/Group | Deep Brain Stimulation(DBS) OFF & ON Medication
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22
PD Phenotype [Count of Participants; unit: Participants]
  Tremor Dominant | 4
  Postural Instability and Gait Disorder(PIGD) | 6
  Intermediate | 12

OUTCOME MEASURES:

1. Primary Outcome: Gait Kinematic Response for 180 and 60Hz DBS
Description: The measurements of interest were captured during the instrumented walk. Interaction of DBS Frequency and Levodopa on gait kinematics was assessed using LM-ANOVA.
Time Frame: 1-2 minute period with each stimulation condition in the Medicated and Unmedicated states.
Population: Scale range 0-100 ( toe angle - higher value is a better outcome; Single limb support - higher value is better outcome; left foot stance % - higher value is worse outcome; left foot swing - higher value is better outcome; left arm range of motion - higher value is better outcome)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- 180HZ (OFF MED): DBS at 180Hz in the OFF Levodopa states
- 180Hz (ON Med): DBS at 180Hz in the On Levodopa state
- 60Hz (OFF Med): DBS at 60Hz in the OFF Levodopa state
- 60Hz (ON MED): DBS at 60Hz in the On Levodopa state
Arm/Group | 180HZ (OFF MED) | 180Hz (ON Med) | 60Hz (OFF Med) | 60Hz (ON MED)
Number analyzed (Participants) | 22 | 22 | 22 | 22
units on a scale
  Right Toe off Angle | 27.37 (1.08) | 29.05 (1.09) | 25.68 (1.08) | 28.31 (1.09)
  Right Single Limb Support | 35.77 (0.56) | 36.44 (0.56) | 35.10 (0.56) | 36.47 (0.56)
  Left Foot Stance | 64.23 (0.55) | 63.48 (0.56) | 64.94 (0.55) | 63.52 (0.56)
  Left Foot Swing | 35.77 (0.55) | 36.52 (0.56) | 35.07 (0.55) | 36.48 (0.56)
  Left Arm Range of Motion | 19.13 (1.94) | 25.37 (1.99) | 17.98 (1.95) | 20.48 (1.98)
Statistical Analysis 1: Comparison: 180HZ (OFF MED) vs 180Hz (ON Med) vs 60Hz (OFF Med); Test type: Other — A linear mixed-effects analysis of variance (LM-ANOVA) model was used to determine the effect of L-Dopa, frequency, the interaction of levodopa and frequency, and the interaction of frequency and contact pairs on gait parameters. The fixed effects were L-Dopa condition (ON vs. OFF), stimulation frequency (LFS;60 Hz vs. HFS;180 Hz), contact pairs [1-(R)/1-(L); 2-(R)/2-(L); 3-(R)/3-(L); 4-(R)/4-(L)], and assistive device (presence vs. absence) and the patient effect was considered random; p < 0.05, Mixed Models Analysis

2. Primary Outcome: Accuracy of Discriminating STN-DBS (60hz vs. High Frequency) and Medication States With Machine Learning(ML)
Description: We apply ML techniques to a data set of gait kinematics acquired from instrumented walking assessments and utilize random forest ML algorithms to identify participants' stimulation frequency/medication condition.
Time Frame: 2 years
Population: The random forest classifier's predictive accuracy for discriminating OFF DBS/OFF MED condition from alternative DBS/MED conditions is listed below.
Measure: Number; unit: percentage of random forest accuracy
Groups:
- Subthalamic-DBS at 60Hz and 180Hz in the Levodopa OFF and ON State.: Deep Brain Stimulation: Each DBS electrode contact was reprogrammed in Low Frequency Stimulation (LFS;60hz) and High Frequency Stimulation (HFS; 180hz) in the Levodopa ON (medicated) and OFF (unmedicated) conditions.
Arm/Group | Subthalamic-DBS at 60Hz and 180Hz in the Levodopa OFF and ON State.
Number analyzed (Participants) | 21
percentage of random forest accuracy | 64

3. Secondary Outcome: Change in Hand Tremor Severity for 180 and 60Hz DBS
Description: The difference in tremor (e.g. rest, postural) severity will be measured with the kinesia sensor for each DBS electrode stimulation pair (60hz or High Frequency) in both the medicated and unmedicated states on a severity scale from 0-4. Higher number = worse outcome
Time Frame: 1 minute test session for each stimulation condition
Population: There was significant difference between rest and postural tremor between 60Hz and 180hz
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- 180Hz DBS (OFF Med): DBS at 180Hz in the OFF Levodopa state
Arm/Group | 180Hz DBS (OFF Med) | 180Hz (ON Med) | 60Hz (OFF Med) | 60Hz (ON Med)
Number analyzed (Participants) | 22 | 22 | 22 | 22
score on a scale
  Left Rest Tremor | 0.19 (0.08) | 0.19 (0.08) | 0.51 (0.08) | 0.40 (0.08)
  Left Hand Postural Tremor | 0.23 (0.09) | 0.13 (0.09) | 0.66 (0.09) | 0.46 (0.09)
  Right Hand Rest Tremor | 0.27 (0.12) | 0.23 (0.11) | 0.57 (0.12) | 0.45 (0.11)
  Right Hand Postural Tremor | 0.22 (0.09) | 0.16 (0.10) | 0.58 (0.10) | 0.42 (0.10)

4. Secondary Outcome: Change in Speed of Limb Movements for 180 and 60Hz DBS
Description: The difference in the speed of limb movements (e.g. hand grasps and leg lifts) will be measured with the kinesia sensor for each DBS electrode stimulation pair (60hz or High Frequency) in both the medicated and unmedicated states on a severity scale of 0-4. Higher values = worse outcome.
Time Frame: 1 minute test session for each stimulation condition
Population: There were no significant difference between groups
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- 180Hz (OFF MED: DBS at 180Hz in the OFF Levodopa state
Arm/Group | 180Hz (OFF MED | 180Hz (ON Med) | 60Hz (OFF Med) | 60Hz (ON Med)
Number analyzed (Participants) | 22 | 22 | 22 | 22
score on a scale
  Left Hand Movement Speed | 2.65 (0.11) | 2.55 (0.11) | 2.76 (0.11) | 2.58 (0.11)
  Right Hand Movement Speed | 2.85 (0.11) | 2.70 (0.11) | 2.90 (0.11) | 2.73 (0.11)

ADVERSE EVENTS:
Time Frame: Adverse events was assessed during each study visit day. At total of 2-3 study visits over 6 weeks
Description: Adverse Events were monitored for all enrolled subjects during the study period.
Groups:
- OFF Medication/OFF DBS: Subthalamic-Deep Brain Stimulation OFF / OFF L-Dopa
- ON Medication/ OFF DBS: Subthalamic- Deep Brain StimulationOFF/ ON L-dopa
- 60Hz DBS (OFF Med): Subthalamic- Deep Brain Stimulation(60hz) and OFF L-Dopa
- 60Hz DBS (ON Med); 180Hz (ON Med): Subthalamic- Deep Brain Stimulation(60hz) and ON L-Dopa
- 180Hz (OFF Med): Subthalamic- Deep Brain Stimulation(180hz) and OFF L-Dopa
Arm/Group | OFF Medication/OFF DBS | ON Medication/ OFF DBS | 60Hz DBS (OFF Med) | 60Hz DBS (ON Med) | 180Hz (OFF Med) | 180Hz (ON Med)
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-12): https://cdn.clinicaltrials.gov/large-docs/91/NCT04184791/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/91/NCT04184791/ICF_001.pdf